CLINICAL TRIAL: NCT02559531
Title: Reliability of the Swiss Emergency Triage Scale (SETS®) Used by Emergency Medical Service (EMS) Providers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Olivier T. Rutschmann, MD, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCER 15-083
Record Dates: First submitted 2015-09-21; First posted 2015-09-24 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Emergency Medical Services; Triage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention group (Experimental): EMS providers will evaluate computerized clinical scenarios using a mobile triage device
  Interventions: Device: Mobile triage system

INTERVENTIONS:
Device: Mobile triage system — A mobile triage system used by EMS providers will be evaluated using standardized clinical vignettes

SUMMARY:
The Swiss Emergency Triage Scale (SETS) in used for triage in emergency departments in Switzerland, France and Belgium. No validated triage scale is actually used by Emergency Medical Service (EMS) providers. The objective of this project is to evaluate the reliability and performance of triage by EMS providers with the SETS.

DETAILED DESCRIPTION:
The Swiss Emergency Triage Scale (SETS) in used for triage in emergency departments in Switzerland, France and Belgium. No validated triage scale is actually used by EMS providers. The objective of this project is to evaluate the reliability and performance of triage by EMS providers with the SETS.

In order to perform this evaluation a cohort of 22 EMS providers will evaluate 28 standardized clinical scenarios using a computer simulator.

ELIGIBILITY:
Inclusion Criteria:

* All EMS providers employed by a private ambulance company in the State of Geneva, Switzerland

Exclusion Criteria:

* Not giving informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Emergency level (1 to 4) accordingly to the SETS | 1 day: all computeriez vignettes will be evaluated during a one-day session in November 2015.
  Each participant will attribute an emergency level (1 to 4) to all clinical vignettes accordingly to SETS criteria. Reliability will be evaluated by computing inter-rater reliability using Kappa statistics.

SECONDARY OUTCOMES:
Correct emergency triage level identification | 1 day: all computeriez vignettes will be evaluated during a one-day session in November 2015.
  Triage levels attributed by EMS providers will be compared with triage levels attributed by experts
Proper orientation | 1 day: all computeriez vignettes will be evaluated during a one-day session in November 2015.
  At the end of triage process, EMS providers have to decide in which hospitals the patients should be admitted. These orientations given by EMS providers will be compared with orientations attributed by experts

CONTACTS AND LOCATIONS:
Overall Officials: Olivier T Rutschmann, MD, MPH, Principal Investigator — University Hospital, Geneva
Locations (1):
- ED of Geneva University Hospitals, Geneva, Canton of Geneva, Switzerland